CLINICAL TRIAL: NCT05114265
Title: A Phase 1 Randomized, Double-Blind, Two Part Study of the Safety, Tolerability, Pharmacokinetics, Analgesic and Respiratory Effect of KUR-101 in Healthy Adult Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of KUR-101 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kures, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KUR-101-101
Record Dates: First submitted 2021-10-19; First posted 2021-11-09 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Single ascending dose (Experimental): Single dose of oral KUR-101 or oral placebo
  Interventions: Drug: KUR-101; Drug: Placebo
- Part 2: Three-way crossover (Experimental): Single dose of oral KUR-101, oral placebo and oral OxyNorm
  Interventions: Drug: KUR-101; Drug: OxyNorm; Drug: Placebo

INTERVENTIONS:
Drug: KUR-101 — Single oral dose of KUR-101
Drug: OxyNorm — Single oral dose of OxyNorm
  Arms: Part 2: Three-way crossover
Drug: Placebo — Single oral dose of placebo

SUMMARY:
This project is testing the safety, tolerability, pharmacokinetics (PK, the amount of study drug in your blood) and pharmacodynamics (PD, how the study drug affects your body) of single doses of a new drug called KUR-101.

Up to 58 healthy men or women aged between 18-55 will be enrolled in this study in two parts.

Part 1 will involve a single ascending (increasing) dose (SAD) where 40 participants (5 groups of 8) will be randomised (assigned randomly, like flipping a coin) to receive a single oral dose of the study drug or placebo. The placebo will look the same as the study drug but will not contain any medicine.

Part 2: will involve a crossover design where 18 participants will be randomised to receive a single oral dose of each of three interventions (study drug, placebo or a marketed form of oxycodone). Each dose is separated by 7 days and the participants are randomised so they do not know the order of the interventions.

For Part 1 the total participation will last 9 days, of which 4 days (3 nights) will be spent in the clinic. One group of subjects in Part 1 will return to the clinic to receive a second dose of drug given with a high fat breakfast. In this group, the total participation will last 16 days, of which 8 days (7 nights) will be spent in the clinic.

For Part 2 the total participation will last 23 days, of which 9 days (8 nights) will be spent in the clinic.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, prospective, study of orally administered KUR-101 in normal healthy participants. The study will be conducted in two parts.

Part 1 is a randomized, double-blind, placebo-controlled study to assess the safety, tolerability, PK, analgesic and respiratory effects of single ascending doses of orally administered KUR-101 in normal healthy participants. Once the MTD has been determined, this dose, or an alternate lower dose, will be taken into Part 2 of the study.

Part 2 is a randomized, double-blind, placebo-controlled, three-period crossover study to assess the analgesic and respiratory effects of a single oral KUR-101 as compared to that of oxycodone in normal healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects;
* Between 18 and 55 years of age;
* Provide a signed EC-approved consent form;
* Generally healthy, in the opinion of the Investigator;
* Body Mass Index (BMI) 18 to 32 kg/m^2;
* Using method of contraception;
* Willing and able to comply with protocol requirements for the duration of the study

Exclusion Criteria:

* Subjects taking prohibited medications;
* Subjects with a history or presence of clinically significant medical or psychiatric disease;
* Subjects with a history of recreational or opiate use;
* Subjects with a history of alcohol abuse or moderate to severe substance abuse;
* Subjects who have regularly used nicotine-containing products;
* Subjects with a hospital admission or major illness within 1 month prior to Screening;
* Subjects with a major surgery within 3 months prior to Screening;
* Subjects who are pregnant or breastfeeding
* Subjects who have participated (taken investigative drug and/or device) in another clinical trial within 30 days prior to Screening;
* Subjects who belong to a vulnerable population.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Part 1: Safety of KUR-101 when compared with placebo | From the signing of the informed consent through Day 8 in Cohort 1, 2, 4 and 5 and through Day 15 in Cohort 3
  Measured by the incidence of treatment-emergent adverse events
Part 2: Effect of KUR-101 on evoked pain response as compared to oxycodone and placebo | Up to 4 hours post dose
  Measured using the cold pressor test
Part 2: Effect of KUR-101 on evoked pain response as compared to oxycodone and placebo | Up to 4 hours post dose
  Measured using thermal sensory testing

SECONDARY OUTCOMES:
Part 1 and Part 2: Pharmacokinetics of KUR-101 | Up to 48 hours post dose
  Measured by levels of KUR-101 in the blood
Part 1: Pharmacokinetics of KUR-101 | Up to 48 hours post dose
  Measured by levels of KUR-101 in the urine
Part 1: Effect of KUR-101 on respiratory function when compared to placebo | Up to 8 hours post dose
  Measured using continuous end-tidal capnography monitoring
Part 1: Effect of KUR-101 on respiratory function when compared to placebo | Up to 8 hours post dose
  Measured using pulse oximetry
Part 1: Effect of KUR-101 on respiratory function when compared to placebo | Up to 8 hours post dose
  Measured using vital signs monitoring
Part 2: Effect of KUR-101 on respiratory function when compared to placebo and oxycodone | Up to 8 hours post dose
  Measured using continuous end-tidal capnography monitoring
Part 2: Effect of KUR-101 on respiratory function when compared to placebo and oxycodone | Up to 8 hours post dose
  Measured using pulse oximetry
Part 2: Effect of KUR-101 on respiratory function when compared to placebo and oxycodone | Up to 8 hours post dose
  Measured using vital signs monitoring
Part 2: Safety of KUR-101 when compared with placebo and oxycodone | From the signing of the informed consent through Day 22
  Measured by the incidence of treatment-emergent adverse events
Part 2: Addictive potential of KUR-101 when compared with placebo and oxycodone | Up to 4 hours post dose
  Measured through the Desire for Opioids visual acuity scale
Part 2: Addictive potential of KUR-101 when compared with placebo and oxycodone | Up to 4 hours post dose
  Measured through the Addiction Research Center Inventory Morphine Benzedrine Group scale

OTHER OUTCOMES:
Part 1: Effect of KUR-101 on evoked pain response as compared to placebo | Day 1 up to 4 hours post dose
  Measured using the cold pressor test
Part 1: Addictive potential of KUR-101 when compared with placebo | Up to 4 hours post dose
  Measured through the Desire for Opioids visual acuity scale
Part 1: Addictive potential of KUR-101 when compared with placebo | Up to 4 hours post dose
  Measured through the Addiction Research Center Inventory Morphine Benzedrine Group scale

CONTACTS AND LOCATIONS:
Locations (1):
- KUR-101-101 Clinical Research Site, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No